CLINICAL TRIAL: NCT06240026
Title: Effects of Transauricular Vagal Nerve Stimulation on Interoceptive Channels in Healthy Subjects
Brief Title: Transauricular Vagal Nerve Stimulation, Pressure Pain and Interoception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Laura De Herde, Principle Investigator, Aalborg University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: N-20230022
Record Dates: First submitted 2024-01-15; First posted 2024-02-02 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Pain, Acute
Keywords: transauricular Vagal Nerve Stimulation; Interoception; Deep Muscular Pressure Pain; Mechanism; Cardioception; Thermoception
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Intervention Model Description: In the first experiment, participants will part-take in two identical stimulation sessions, differing only by the use of active taVNS in one session and an active control of left earlobe stimulation in the other. The sequence of sessions will be counter-balanced and randomized between participants.
  In the second experiment, participants will part-take in two sessions, occurring on 2 different days separated by 48h minimum. In each session, participants will undergo three 40 min stimulation, separated by 30min and differing in location, intensity and paradigm. Specifically, in one session, participants will undergo taVNS-burst-high-intensity, taVNS-continuous-high-intensity and taVNS-continuous-low-intensity (randomized). In the second session, participants will undergo earlobe-burst-high-intensity, earlobe-continuous-high-intensity and sham (in the complementary order to the other session). The sequence of sessions will be counter-balanced and randomized between participants.
Who Masked: Participant, Investigator
Masking Description: Electrodes for taVNS and earlobe stimulation will be placed onto the participant during both stimulation sessions. These electrodes have identical wires which are connected to a digitimer for the control of the stimulation.
  Researchers doing the stimulation will have no other role in the study and will not participate in patient assessment.
  Participants will be blinded to which stimulation type is termed 'taVNS'. And only individuals having no prior experience with taVNS will be recruited. Care will be taken not to set research appointments with participants close one to the others to avoid waiting room conversations between participants. Efficacy of blinding will be assessed at the end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- transauricular Vagal Nerve Stimulation (Experimental): NEMOS taVNS electrodes will be placed in the left concha cymba of participants (CerboMed GmbH, Erlangen, Germany). When appropriate, these electrodes will be plugged into a digitimer. Whilst pulse width, frequency, stimulation burst and total duration will be respectively standardized to 200microseconds and 25Hz.
  In the first experiment, continuous and 20min stimulation will be applied at one person-specific intensity. To acquire this, using an elegant stair-case algorithm, perception and supra-pain (described as a 7/10 pain level, where 10 is the most amount of pain imaginable) thresholds will be obtained. Stimulation intensity will then be defined as 2/3 the range between these thresholds.
  In the second experiment, burst and continuous stimulation will be applied for 40min. Two intensities will be used: 2/3 the range between perception and supra-pain thresholds and supra-pain thresholds.
  Interventions: Device: taVNS
- Earlobe Stimulation (Active Comparator): Electrodes (Ambu, Neuroline, Bordeaux, France) will respectively be placed on the front and back of the earlobe. When appropriate, these electrodes will be plugged into a digitimer . Whilst pulse width, frequency, stimulation burst and total duration will be respectively standardized to 200microseconds, 25Hz, continuous and 20minutes, the stimulation will be person specific. To acquire this intensity, participants will perform a thresholding protocol. Based on an elegant stair-case algorithm, the perception and pain (described as a 7/10 pain level, where 10 is the most amount of pain imaginable) thresholds will be obtained. Stimulation intensity will then be defined as 2/3 the range between these thresholds. For example, if the perception and pain thresholds are respectively at 2mA and 8mA, the stimulation intensity would be 6mA.
  Interventions: Device: Earlobe Stimulation
- Sham (Sham Comparator): No current will be applied to the ear of the participant.
  Interventions: Device: taVNS; Device: Earlobe Stimulation

INTERVENTIONS:
Device: taVNS — transauricular vagal nerve stimulation electrodes (NEMOS, CerboMed GmbH, Erlangen, Germany), attached to a digitimer.
  Arms: Sham; transauricular Vagal Nerve Stimulation
Device: Earlobe Stimulation — Standard electrodes (Ambu, Neuroline, Bordeaux, France) cut into 0.6cm circles, attached to a digitimer.
  Arms: Earlobe Stimulation; Sham

SUMMARY:
Interoception, the ability to perceive, process and respond to signals originating from within the body, is crucial for maintaining healthy physiological ranges. Indeed, dysfunction in this ability has been associated with various mood and pain disorders. Based on the overlap between the anatomical pathway of this ability and the site of action of the tool, transauricular vagal nerve stimulation (taVNS) could modulate this interoception. However, little is known about the breadth, duration, and mechanism of interoception modulation by taVNS.

The study (Ethics Region Nord Jylland Denmark, N-20230022) will address these limitations, with 2 experiments with a focus on three interoceptive channels: deep muscular pressure pain, heartbeat, and thermal perception.

DETAILED DESCRIPTION:
The first experiment will aim to corroborate and extend the pain-modulating effect of taVNS to other interoceptive functions and to vagal-activation markers. For this, 30 healthy subjects will complete a randomized, active control, crossover study. The main intervention is left concha taVNS (NEMOS, CerboMed GmbH, Erlangen, Germany) for 20 minutes (200µs duration, 25Hz, at a personalized intensity). This will be compared to an active control of identical electrical stimulation to the left earlobe. A blinding assessment inquiring which stimulation is supposed to be therapeutic will be collected. Main outcomes are pressure pain thresholds and temporal summation of pain responses acquired via cuff-pressure algometer (Cortex Technology, Aalborg University, Denmark) placed at the calf. Heartbeat perception, assessed via the heartbeat counting task, and thermal perception, assessed using a QST thermal grid, are also primary outcomes. Secondary outcomes are conditioned pain modulation, resting state electroencephalography, electrocardiography, and pupillary light reflexes. To assess whether, and how, taVNS modulates deep muscular pressure pain, heartbeat, and thermal perception, primary and secondary measurements pre, post and 30min post stimulation will be collected and compared. To assess the duration of the potential effects, these outcomes will be collected, and compared, at 5min intervals until the primary measurements are within 20% of baseline values. Given baseline is recovered, the second stimulation session will take place. Given this has not occurred within 1.5h of the cessation of the stimulation in the first stimulation session, subjects will be asked to come back at their earliest convenience.

The second experiment will additionally explore the effect of stimulation paradigm and intensity. For this, 20 healthy subjects will complete a randomized, active and sham control, crossover study. The main intervention is left concha taVNS (NEMOS, CerboMed GmbH, Erlangen, Germany) for 40 minutes (200µs duration, 25Hz). This will be compared to an active control of identical electrical stimulation to the left earlobe and sham stimulation. Stimulation intensity will be given at 2/3rd of perception to pain threshold and at pain thresholds. A burst and continuous paradigm will also be employed. A blinding assessment inquiring which stimulation is supposed to be therapeutic will be collected. Main outcomes are pressure pain thresholds acquired via cuff-pressure algometer (Cortex Technology, Aalborg University, Denmark) placed at the calf. Heartbeat perception, assessed via the heartbeat counting task is also primary outcomes. Secondary outcomes are conditioned pain modulation, resting state electroencephalography, electrocardiography, and pupillary light reflexes. Assessments will be acquire pre, during and post stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Are aged 18-60
* Are healthy
* Speak and understand English

Exclusion Criteria:

* Are pregnant and/or breastfeeding
* Regularly use cannabis, opioids, or other drugs
* Currently or previously suffered of a neurologic, musculoskeletal, mental, or other illnesses (e.g., brain or spinal cord injuries, degenerative neurological disorders, major depression, cardiovascular disease, chronic lung disease, etc.)
* Once or more a week take of analgesic medication or other medication which may affect the trial (including paracetamol and NSAIDs)
* Have a recent history of acute pain, particularly in the lower limbs.
* Have abnormally disrupted sleep in 24 hours preceding experiment.
* Have contraindications to electric application (history of epilepsy, metal implants in head or jaw, etc.)
* Lack the ability to cooperate.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-08-07 (Actual); Study Completion 2025-08-07 (Actual)

PRIMARY OUTCOMES:
Pain Perception Threshold | This measurement will be taken pre-intervention, and directly post- and 30min post-intervention. It will also be taken in 5min intervals post-intervention until the PPT is back within 20% of the pre-intervention value.
  Pressure algometer cuffs, placed on the calf of participants, attached to an electronic visual analogue scale (VAS) measuring device will be employed. Per cuff, as it inflates, participants are asked to move the dial of the VAS when the pressure begins to be painful. The pressure at which this occurs is referred to as the pain perception threshold (PPT).
Pain Tolerance Threshold | This measurement will be taken pre-intervention, and directly post- and 30min post-intervention.
  Pressure algometer cuffs, placed on the calf of participants, attached to a visual analogue scale (VAS) will be employed. Per cuff, as it inflates, participants are asked to move the dial of the VAS when the pressure begins to be painful. They are then tasked to accordingly move the dial as the pain increases. Importantly, when the pain becomes intolerable, participants are tasked to press the red button which releases all pressure. The pressure at which this occurs is referred to as the pain tolerance threshold (PTT).
Temporary Summation of Pain | This measurement will be taken pre-intervention, and directly post- and 30min post-intervention.
  The pressure algometer cuff will inflate on the dominant leg for 1second, with a 1second break, to the given PTT 10 times consecutively. Participants are asked to move the VAS dial to the pain level at each inflation, without returning to 0 on the scale. Nothing will be done with the cuff on the opposite leg.
Heartbeat Perception | This measurement will be taken pre-intervention, and directly post- and 30min post-intervention.
  Randomly interleaved and without manual help, subjects will be tasked to count their own heartbeat across 3 time-intervals (25, 35 and 45 seconds). The difference between the perceived and actual heartbeat count is defined herein as the heartbeat perception.
Thermal Perception | This measurement will be acquired pre-intervention, and directly post- and 30min post-intervention.
  The QST.lab thermal stimulator contains 6 stimulation regions, which can individually be programmed. First, with all regions programmed identically, participants will be tasked to state when the stimulus is perceived as painfully cold and warm. These will respectively be the cold and warm thresholds. A thermal-grid illusion pattern will then be generated: this involves interleaving stimulation regions as cold (2deg above the cold threshold) and hot (2deg below the hot threshold). Participants will then be asked to rate the pain intensity of this stimulation (0=no pain, 10=worst pain imaginable).

SECONDARY OUTCOMES:
Conditioned Pain Modulation | This measurement will be taken pre-intervention, and directly post- and 30min post-intervention.
  The non-dominant leg will receive a continuous pressure of 70% of the PTT previously registered. The cuff on the dominant leg will gradually inflate. As this occurs, participants are once again asked to start moving the dial when the pressure begins to be painful, and to press the red button when this becomes intolerable.
Handheld Pain Perception Threshold | This measurement will be taken pre-intervention, and directly post- and 30min post-intervention.
  For each side separately, a handheld pressure algometer will be applied at a constant rate of 30kPa/s, perpendicularly to the belly of the musculus trapezius. Participants will be instructed to press a button when they first perceive the pressure to be painful. This is referred to as the handheld pain perception threshold.

OTHER OUTCOMES:
Pupil Light Reflex | This measurement will be taken pre-intervention, and directly post- and 30min post-intervention.
  Using a pupilometer, covering the other eye, the size of one pupil will be measured during the light reflex. This will be done for both eyes.
Resting State Electroencephalography | This measurement will be taken pre-intervention, during the intervention and post- and 30min post-intervention.
  Using electroencephalography (g.tec medical engineering, Austria), namely a cap of electrodes conducted to the head using gel, resting state brain activity will be recorded
Resting State Electrocardiography | This measurement will be taken pre-intervention, and directly post- and 30min post-intervention.
  Using electrocardiography, namely electrodes placed on the torso of participants, resting state cardiac activity will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Neuroplasticity and Pain, Gistrup, North Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No
Data will be anonymized. During the experiment, personal data necessary for the execution of the project will be processed, and after termination of the experiment, personal data in accordance with the Data Protection Regulation.